CLINICAL TRIAL: NCT06855082
Title: A Study of Using the Stoma Self-care Apps by Patients With Enterostomy on the Integrated Model of Technology Acceptance (TAM) and Task-technology Fit(TTF)
Brief Title: A Study of Using the Stoma Self-care Apps by Patients With Enterostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HSIN LING CHEN (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, HSIN LING CHEN, Surgical Ward RN, Mackay Memorial Hospital
Organization: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24MMHIS457e
Record Dates: First submitted 2025-02-14; First posted 2025-03-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Enterostomy
Keywords: Enterostomy; stoma self-care apps; Technology Acceptance Model; Task Technology Fit Model
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Technology Acceptance Model, TAM Task Technology Fit Model, TTF
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stoma self-care apps (Experimental): uses a stoma self-care app, accessed through LINE official account, a communication software commonly used by Chinese people, as an intervention measure to integrate technology acceptance and task technology adaptation models to explore the correlation of each aspect and its impact on self-care ability and quality of life.
  Interventions: Behavioral: stoma self-care apps
- conventional (Placebo Comparator): conventional Traditional Education
  Interventions: Behavioral: Traditional Education Receive colostomy health education manual with oral instruction

INTERVENTIONS:
Behavioral: stoma self-care apps — This study uses a stoma self-care app, accessed through LINE official account, a communication software commonly used by Chinese people, as an intervention measure to integrate technology acceptance and task technology adaptation models to explore the correlation of each aspect and its impact on self-care ability and quality of life. Whether the factors and task technology adaptability will affect the willingness and usage behavior of enterostomy patients, the research subjects can effectively improve their self-care ability, quality of life, usage willingness, and usage behavior after intervention.
  Arms: stoma self-care apps
Behavioral: Traditional Education Receive colostomy health education manual with oral instruction — conventional
  Arms: conventional

SUMMARY:
This study uses a stoma self-care app, accessed through LINE official account, a communication software commonly used by Chinese people, as an intervention measure to integrate technology acceptance and task technology adaptation models to explore the correlation of each aspect and its impact on self-care ability and quality of life. Whether the factors and task technology adaptability will affect the willingness and usage behavior of enterostomy patients, the research subjects can effectively improve their self-care ability, quality of life, usage willingness, and usage behavior after intervention.

DETAILED DESCRIPTION:
Background: Self-care for patients after enterostomy surgery includes both cognitive and skill aspects. Insufficient self-care ability, inability to tell self-care precautions, and incorrect steps in performing care skills lead to leakage of the ostomy bag, and 70% of peristomal skin lesions occur. Complications lead to increased hospitalization days, readmission rates, and medical costs. Pain and other discomforts caused by skin complications around the stoma can cause anxiety, depression or anger, followed by financial burdens and impacts on families, affecting the quality of life. Ostomates use paper texts and oral instructions to provide post-enterostomy nursing care instructions. There is no regular follow-up mechanism after discharge. After returning home, enterostomy patients' self-care ability and adaptability to the stoma will be tested. Changes in the defecation outlet after enterostomy surgery affect many aspects. Patients need to relearn daily care. Physically, they need to maintain the cleanliness of the ostomy bag collection system at all times. Their lifestyle must be consistent with postoperative diet and exercise. Changes; psychologically, the changes in body function and appearance, anxiety, depression, or anger caused in the process of adapting to the enterostomy lifestyle, followed by the financial burden and impact on the family, and the physical, mental, and spiritual impact of family members on each other. It is a huge change, providing ongoing care guidance and support to ensure self-care and quality of life after returning home, meeting the constraints faced by patients with enterostomy needs and the challenges faced by their care guidance.

Purpose: This study uses a stoma self-care app, accessed through LINE official account, a communication software commonly used by Chinese people, as an intervention measure to integrate technology acceptance and task technology adaptation models to explore the correlation of each aspect and its impact on self-care ability and quality of life. Whether the factors and task technology adaptability will affect the willingness and usage behavior of enterostomy patients, the research subjects can effectively improve their self-care ability, quality of life, usage willingness, and usage behavior after intervention.

Method: It is a quantitative, single-blind, simple randomly assigned, quasi-experimental study. The surgical ward and stoma treatment room of a medical center in northern Taiwan accepted patients with enterostomy, including 25 patients in the control group and 25 patients in the experimental group. The interventional measures were performed on the first day after enterostomy surgery, using integrated technology to receive and adapt task technology. Model, the enterostomy self-care knowledge scale, and the stoma self-care ability scale (UES) are used to evaluate self-care ability, and the stoma patient quality of life scale (Stoma-QOL) is used to evaluate the quality of life, and a questionnaire survey is conducted. Analyze task technology fit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer or intestinal obstruction or abdominal trauma, those who have received colostomy during this hospitalization
* Conscious, can communicate in Mandarin or Minnan dialect
* Have no communication, vision, or hearing impairments,
* Have smartphones

Exclusion Criteria:

* Those who are unable to cooperate due to visual, hearing, cognitive or mental impairments
* Patients who need colostomy surgery due to non-colorectal cancer, intestinal obstruction, or abdominal trauma
* Patients diagnosed by a physician as having surgery-related complications and requiring further surgery, such as infection, intestinal Perforation, stoma prolapse, stenosis, necrosis, bleeding, etc. (IV) Those who are unable to learn self-care on the day before discharge due to worsening of their illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
The quality of life of patients with colostomy | Day 1 to 28 after colostomy surgery
  The Stoma-QOL scale was used to measure the quality of life. The score was scored on a 4-point scale ranging from 30 to 120 points. The higher the score, the better the quality of life of the research subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins L, Down G, Andersen BD, Nielsen LF, Hansen AS, Herschend NO, Storling Z. The Ostomy Skin Tool 2.0: a new instrument for assessing peristomal skin changes. Br J Nurs. 2022 Apr 21;31(8):442-450. doi: 10.12968/bjon.2022.31.8.442. PMID 35439075